CLINICAL TRIAL: NCT03003156
Title: 50 Hz vs. 25 Hz Magnetic Seizure Therapy for Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHDC12014111a
Record Dates: First submitted 2016-12-16; First posted 2016-12-26 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Schizophrenia
Keywords: magnetic seizure therapy; schizophrenia; controlled trial; cognition
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 25 Hz magnetic seizure therapy (Experimental): 10 treatment sessions of 25 Hz MST, three times per week in the first two weeks, two times per in the following two weeks.
  Interventions: Procedure: 25 Hz magnetic seizure therapy
- 50 Hz magnetic seizure therapy (Experimental): 10 treatment sessions of 50 Hz MST, three times per week in the first two weeks, two times per in the following two weeks.
  Interventions: Procedure: 50 Hz magnetic seizure therapy

INTERVENTIONS:
Procedure: 25 Hz magnetic seizure therapy — In addition to treatment as usual (TAU), participants were supposed to receive ten sessions of 25 Hz MST in four weeks, with three sessions per week in the first two weeks and two sessions per week in the following two weeks.
  Arms: 25 Hz magnetic seizure therapy
Procedure: 50 Hz magnetic seizure therapy — In addition to treatment as usual (TAU), participants were supposed to receive ten sessions of 50 Hz MST in four weeks, with three sessions per week in the first two weeks and two sessions per week in the following two weeks.
  Arms: 50 Hz magnetic seizure therapy

SUMMARY:
This trial attempts to investigate whether the dosage (frequency) has an effect on the treatment efficacy and cognitive outcomes of magnetic seizure therapy (MST) among schizophrenia patients. Half of the participants will be recruited to receive 25 Hz MST, while the other half will be recruited to 50 Hz MST.

DETAILED DESCRIPTION:
Magnetic seizure therapy (MST) is likely to be an alternative options to electroconvulsive therapy (ECT).Widespread stimulation of cortical and subcortical regions is inevitable for ECT since the substantial impedance of the scalp and skull shuts most of the electrical stimulus away from the brain. Nevertheless, magnetic pulses are capable to focus the stimulus to a specific area of the brain because they can pass the scalp and skull without resistance. In Addition, electric current will penetrate into deeper structures, while magnetic stimulus are only capable to reach a depth of a few centimeters. As a consequence, MST are able to generate focus stimuli on superficial regions of the cortex while ECT can't, which may give MST the capability to produce comparable therapeutic benefits with the absence of apparent cognitive side effects. Though high dose (frequency) MST is gaining popularity, there is no evidences supporting its superiority over low dose (frequency) MST either on efficacy, safety, or seizure quality.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-5 diagnosis of schizophrenia;
2. convulsive therapy clinically indicated, such as severe psychomotor excitement or retardation, attempts of suicide, being highly aggressive, pharmacotherapy intolerance, and ineffectiveness of antipsychotics;
3. the positive and negative syndrome scale (PANSS)[20] score ≥ 60;
4. informed consent in written form.

Exclusion Criteria:

1. diagnosis of other mental disorders;
2. severe physical diseases, such as stroke, heart failure, liver failure, neoplasm, and immune deficiency;
3. present with a laboratory abnormality that could impact on efficacy of treatments or safety of participants;
4. failure to respond to an adequate trial of ECT lifetime;
5. are pregnant or intend to get pregnant during the study;
6. other conditions that investigators consider to be inappropriate to participate in this trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
changes of The Positive and Negative Syndrome Scale (PANSS) | At baseline, 4-week follow-up

SECONDARY OUTCOMES:
changes of The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | At baseline and 4-week follow-up
seizure duration | at each treatment session, up to 4 weeks
Adverse events | up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chunbo Li, PHD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD data